CLINICAL TRIAL: NCT02417233
Title: Improving Engagement to HIV Prevention and Care in North West, South Africa
Brief Title: Engagement to Care South Africa
Acronym: ICARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-10482; P0054377 (Other Grant/Funding Number: PHS Health Resources & Services Admin.)
Record Dates: First submitted 2014-12-12; First posted 2015-04-15 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-11

CONDITIONS: HIV
Keywords: HIV-positive; adherence; engagement to care; mobile Health (mHealth); SMS; peer navigation; retention
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (No Intervention): Participants are administered baseline, 6 month, and 12 month questionnaires and provided with the study incentive (mobile phone airtime) only. This group will not receive any additional engagement to care intervention.
- SMS text message (Active Comparator): Participants are administered baseline, 6 month, and 12 month questionnaires and provided with the study incentive (mobile phone airtime). In addition, they receive automated bi-weekly behavioral text messages aimed at improving health and reducing transmission risk and also automated bi-weekly "check-in" text messages that will trigger a phone call from clinic staff if the participant reports not being well.
  Interventions: Behavioral: SMS text message
- SMS text message + Peer Navigation (Active Comparator): Participants are administered baseline, 6 month, and 12 month questionnaires and provided with the study incentive (mobile phone airtime). In addition, they receive automated bi-weekly behavioral text messages aimed at improving health and reducing transmission risk and also bi-weekly contact from an HIV-positive peer who provides personalized support and with health or other service systems navigation assistance.
  Interventions: Behavioral: SMS text message + Peer Navigation

INTERVENTIONS:
Behavioral: SMS text message — bi-weekly behavioral messages and bi-weekly check-in messages
  Arms: SMS text message
Behavioral: SMS text message + Peer Navigation — bi-weekly behavioral messages plus personalized peer navigation
  Arms: SMS text message + Peer Navigation

SUMMARY:
This study will evaluate the efficacy of two strategies for enhancing overall preventive behaviors, retention in HIV care, and adherence to medication for HIV positive individuals in South Africa: short message service (SMS) text messaging and peer navigation services.

DETAILED DESCRIPTION:
Treatment-as-prevention represents a game changing potential to stem further HIV transmission by ensuring that infected individuals are tested, linked to care, retained in care, and adherent to their regimens. Little is known, however, about the most feasible and cost-effective means to promote overall engagement in care coupled with behavioral risk reduction for HIV positive individuals in South Africa. For this reason, the study proposes to first assess what engagement in care activities are underway in select clinics in the Bojanala Platinum District, North West Province, South Africa, and will then implement and evaluate the feasibility, acceptability, and potential efficacy of two strategies for enhancing overall preventive behaviors, retention in HIV care and adherence to medication. The first strategy will employ automated text message reminders to encourage patients to return for needed care, adhere to their antiretroviral therapy (ART) regimens, and practice safer sex and other risk reduction behaviors. This approach also includes designation of a retention, adherence, and prevention monitor to supervise the system. A second strategy builds on the first model, including the automated text message system, but also utilizes peer navigator-provider teams to serve as point people for care engagement. Peer navigators will work with providers to introduce patients to care and help them establish a care and prevention plan. They will also check in with patients to discuss and support resolution of challenges to engaging in care, adhering to drug regimens, and reducing transmission risk behavior.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive (diagnosed within the last 12 months prior to study/patient contact)
* Has access to a mobile phone
* Willing to receive and respond to text messages and calls from clinic and study staff (all arms)
* Willing to communicate and meet with PN (PN arm)
* Willing to meet with study staff for survey at study start, 6 months, and 12 months (all arms)
* regard study clinic area as the regular clinic for accessing healthcare

Exclusion Criteria:

* First tested positive over 12 months prior to recruitment
* Under the age of 18
* Unable to give informed consent
* Unable to read basic English and with no one to read study sms to participant
* Principally accesses care through a clinic not in the study
* Planning to permanently move away from the area served by the clinic within next 6 months (following enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheri Lippman, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- South Africa (2):
  - Moses Kotane Sub-district clinics, Mabeskraal, Northwest
  - Rustenburg Sub-district clinics, Rustenburg, Northwest

REFERENCES:
- [Derived] Leslie HH, Mooney AC, Gilmore HJ, Agnew E, Grignon JS, deKadt J, Shade SB, Ratlhagana MJ, Sumitani J, Barnhart S, Steward WT, Lippman SA. Prevalence, motivation, and outcomes of clinic transfer in a clinical cohort of people living with HIV in North West Province, South Africa. BMC Health Serv Res. 2022 Dec 26;22(1):1584. doi: 10.1186/s12913-022-08962-8. PMID 36572869
- [Derived] Lippman SA, de Kadt J, Ratlhagana MJ, Agnew E, Gilmore H, Sumitani J, Grignon J, Gutin SA, Shade SB, Gilvydis JM, Tumbo J, Barnhart S, Steward WT. Impact of short message service and peer navigation on linkage to care and antiretroviral therapy initiation in South Africa. AIDS. 2023 Mar 15;37(4):647-657. doi: 10.1097/QAD.0000000000003453. Epub 2022 Dec 5. PMID 36468499
- [Derived] Steward WT, Agnew E, de Kadt J, Ratlhagana MJ, Sumitani J, Gilmore HJ, Grignon J, Shade SB, Tumbo J, Barnhart S, Lippman SA. Impact of SMS and peer navigation on retention in HIV care among adults in South Africa: results of a three-arm cluster randomized controlled trial. J Int AIDS Soc. 2021 Aug;24(8):e25774. doi: 10.1002/jia2.25774. PMID 34435440
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Lippman SA, Shade SB, Sumitani J, DeKadt J, Gilvydis JM, Ratlhagana MJ, Grignon J, Tumbo J, Gilmore H, Agnew E, Saberi P, Barnhart S, Steward WT. Evaluation of short message service and peer navigation to improve engagement in HIV care in South Africa: study protocol for a three-arm cluster randomized controlled trial. Trials. 2016 Feb 6;17:68. doi: 10.1186/s13063-016-1190-y. PMID 26852237

RESULTS

PARTICIPANT FLOW:
Groups:
- Short Message Service (SMS) Text Message: Participants are administered baseline, 6 month, and 12 month questionnaires and provided with the study incentive (mobile phone airtime). In addition, they receive automated bi-weekly behavioral text messages aimed at improving health and reducing transmission risk and also automated bi-weekly "check-in" text messages that will trigger a phone call from clinic staff if the participant reports not being well.
  SMS text message: bi-weekly behavioral messages and bi-weekly check-in messages
- Short Message Service (SMS) Text Message + Peer Navigation: Participants are administered baseline, 6 month, and 12 month questionnaires and provided with the study incentive (mobile phone airtime). In addition, they receive automated bi-weekly behavioral text messages aimed at improving health and reducing transmission risk and also bi-weekly contact from an HIV-positive peer who provides personalized support and with health or other service systems navigation assistance.
  SMS text message + Peer Navigation: bi-weekly behavioral messages plus personalized peer navigation
Period: Overall Study
Arm/Group | Standard of Care | Short Message Service (SMS) Text Message | Short Message Service (SMS) Text Message + Peer Navigation
Started | 169 | 289 | 298
Completed | 133 | 238 | 239
Not Completed | 36 | 51 | 59
Not completed — Death | 4 | 10 | 14
Not completed — Lost to Follow-up | 27 | 39 | 34
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 8
Not completed — Relocation out of study area | 1 | 0 | 1
Not completed — Mentally unstable | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 2 duplicate participants and 2 participants who were later found not to be HIV+ (not eligible) were removed from analysis. The first participant who was not HIV+ was dishonest about their status; the second person who was not HIV+ had a reactive rapid test but the confirmatory Western Blot was negative.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | SMS Text Message | SMS Text Message + Peer Navigation | Total
Number analyzed (Participants) | 167 | 289 | 296 | 752
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 167 | 289 | 294 | 750
  >=65 years | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 116 | 106 | 292
  Male | 97 | 173 | 190 | 460
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 166 | 288 | 295 | 749
  Colored | 1 | 0 | 1 | 2
  Missing | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Linkage to Care - Participants Who Received Cluster of Differentiation 4 (CD4) T-cell Count Test Result Within 3 Months of Testing HIV-positive (Binary)
Description: Participants who received CD4 count test result within 3 months of testing HIV-positive (binary)
Time Frame: 3 months
Population: Analysis population is participants who were newly diagnosed HIV+ within 7 days of study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Short Message Service (SMS) Text Message | SMS Text Message + Peer Navigation
Number analyzed (Participants) | 87 | 132 | 133
Participants | 80 | 121 | 119
Statistical Analysis 1: Comparison: Standard of Care vs Short Message Service (SMS) Text Message; Test type: Other; p = 0.848, Regression, Logistic; Odds Ratio (OR) = 0.958, 95% CI 2-sided [0.62 to 1.49]
Statistical Analysis 2: Comparison: Standard of Care vs SMS Text Message + Peer Navigation; Test type: Other; p = 0.125, Regression, Logistic; Odds Ratio (OR) = 1.492, 95% CI 2-sided [0.90 to 2.49]

2. Primary Outcome: Timely Antiretroviral Therapy (ART) Initiation (Participants Eligible for ART Who Initiate Treatment Within 3 Months of Diagnosis)
Description: Participants eligible for ART who initiate treatment within 3 months of diagnosis
Time Frame: 3 months
Population: Analysis population is participants who were newly diagnosed HIV+ within 7 days of study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | SMS Text Message | SMS Text Message + Peer Navigation
Number analyzed (Participants) | 87 | 132 | 133
Participants | 55 | 79 | 94
Statistical Analysis 1: Comparison: Standard of Care vs SMS Text Message; Test type: Other; p = 0.636, Regression, Logistic; Odds Ratio (OR) = 0.866, 96% CI 2-sided [0.48 to 1.57]
Statistical Analysis 2: Comparison: Standard of Care vs SMS Text Message + Peer Navigation; Test type: Other; p = 0.165, Regression, Logistic; Odds Ratio (OR) = 1.401, 95% CI 2-sided [0.87 to 2.26]

3. Primary Outcome: Retention in Care - ART Eligible (Participants Eligible for ART Who Initiated ART and Who Remain on Treatment)
Description: Participants eligible for ART who initiated ART and who remain on treatment 12 months from enrollment. Retention in care at 12 months is defined as at least 4 clinical care visits with less than 4 months between each visit.
Time Frame: 12 months
Population: Analysis population is all enrolled participants who were prescribed ART.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | SMS Text Message | SMS Text Message + Peer Navigation
Number analyzed (Participants) | 139 | 234 | 255
Participants | 77 | 153 | 178
Statistical Analysis 1: Comparison: Standard of Care vs SMS Text Message; Test type: Other; p = 0.16, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.86 to 2.55]
Statistical Analysis 2: Comparison: Standard of Care vs SMS Text Message + Peer Navigation; Test type: Other; p = 0.03, Regression, Logistic; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.06 to 3.14]

4. Primary Outcome: Retention in Care - Non-ART (Participants Who Return for Repeat CD4 Testing Within 12 Months of Diagnosis)
Description: Participants who return for repeat CD4 testing within 12 months of diagnosis
Time Frame: 12 months
Population: Analysis population is all enrolled participants who were not prescribed ART
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | SMS Text Message | SMS Text Message + Peer Navigation
Number analyzed (Participants) | 28 | 55 | 41
Participants | 3 | 2 | 11
Statistical Analysis 1: Comparison: Standard of Care vs SMS Text Message; Test type: Other; p = 0.24, Regression, Logistic; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.03 to 2.45]
Statistical Analysis 2: Comparison: Standard of Care vs SMS Text Message + Peer Navigation; Test type: Other; p = 0.20, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [0.59 to 12.16]

5. Primary Outcome: Adherence to ART - Objective (Viral Load Test Results <400 Copies/mL)
Description: Viral load test results <400 copies/mL (consistent with current and correct adherence to ART)
Time Frame: 12 months
Population: Analysis population is all enrolled participants who were prescribed ART and had received viral load testing by 12 months of study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | SMS Text Message | SMS Text Message + Peer Navigation
Number analyzed (Participants) | 76 | 157 | 160
Participants | 67 | 141 | 132
Statistical Analysis 1: Comparison: Standard of Care vs SMS Text Message; Test type: Other; p = 0.093, Regression, Logistic; Odds Ratio (OR) = 1.943, 95% CI 2-sided [0.90 to 4.21]
Statistical Analysis 2: Comparison: Standard of Care vs SMS Text Message + Peer Navigation; Test type: Other; p = 0.152, Regression, Logistic; Odds Ratio (OR) = 1.764, 95% CI 2-sided [0.81 to 3.83]

6. Primary Outcome: Adherence to ART - Subjective (Self-reported Ability to Take ART as Prescribed in Last Month)
Description: Self-reported ability to take ART as prescribed in last month, assessed at 12 months from enrollment. Considered compliant if reported "very good" or "excellent" adherence.
Time Frame: 12 months
Population: Analysis population is all enrolled participants prescribed ART who returned to answer the 12 month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | SMS Text Message | SMS Text Message + Peer Navigation
Number analyzed (Participants) | 115 | 201 | 214
Participants | 92 | 130 | 162

ADVERSE EVENTS:
Time Frame: "0 participants at risk" included because: Serious and Other Adverse Events were not monitored/assessed in this study because it was not a clinical trial of a new drug or device, but rather, a behavioral intervention. Study staff were not clinicians - only data monitoring assistants and peer health navigators. The study was based in a public clinic system, but the only clinical data abstracted for the study was for the study outcomes described. Other medical data was not recorded.
Description: "0 participants at risk" included because: Serious and Other Adverse Events were not monitored/assessed in this study because it was not a clinical trial of a new drug or device, but rather, a behavioral intervention. Study staff were not clinicians - only data monitoring assistants and peer health navigators. The study was based in a public clinic system, but the only clinical data abstracted for the study was for the study outcomes described. Other medical data was not recorded.
Arm/Group | Standard of Care | SMS Text Message | SMS Text Message + Peer Navigation
All-Cause Mortality (participants affected / at risk) | 4/169 | 10/289 | 14/298
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No